CLINICAL TRIAL: NCT03655041
Title: 24-Weeks of β-Alanine Ingestion on Muscle Taurine and Clinical Blood Parameters in Healthy Males
Brief Title: 24-Wk β-Alanine Ingestion on Muscle Taurine and Clinical Blood Parameters in Healthy Males
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Bruno Gualano, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 24WKBA
Record Dates: First submitted 2018-08-28; First posted 2018-08-31 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Sports Nutritional Physiological Phenomena
Keywords: Physiological Phenomena
MeSH Terms: interventions — beta-Alanine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beta-Alanine (Experimental): 6.4 g/day of beta-alanine for 24 weeks
  Interventions: Dietary Supplement: Beta-alanine
- Placebo (Placebo Comparator): 6.4 g/day of maltodextrin for 24 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Beta-alanine — Beta-alanine in sustained-release tablets to increase muscle carnosine content
  Arms: Beta-Alanine
Dietary Supplement: Placebo — Maltodextrin is used as a placebo as it does not lead to any increases in muscle carnosine
  Arms: Placebo

SUMMARY:
Although β-alanine (BA) has been shown to be an effective ergogenic aid, little information exists on the safety of chronic supplementation despite potential concerns. The aim of this study was to investigate the effects of chronic BA supplementation on muscle taurine content, blood clinical markers and sensory side-effects during 24 weeks of BA supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males

Exclusion Criteria:

* Smokers
* Chronic disease
* Prior or current use of steroids
* Use of creatine in the last 6 months
* Use of beta-alanine in the last 6 months

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2013-02-01 (Actual); Primary Completion 2015-12-15 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
Muscle taurine content in mmol/kg | Up to 24 weeks
  Change in the content of taurine in muscle will be determined using High-Pressure Liquid Chromatography of muscle biopsies

SECONDARY OUTCOMES:
Aspartate transaminase; alanine aminotransferase; alkaline phosphatase; lactate dehydrogenase and creatine kinase in U/L | Up to 24 weeks
  Aspartate transaminase; alanine aminotransferase; alkaline phosphatase; lactate dehydrogenase and creatine kinase will be analysed from venous blood samples
Albumin; globulin; creatinine in mg/dL | Up to 24 weeks
  Albumin; globulin; creatinine will be analysed from venous blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Gualano, PhD, Principal Investigator — University of Sao Paulo

IPD SHARING:
Plan to Share IPD: No